CLINICAL TRIAL: NCT02301208
Title: A Randomized Phase III Study of Concurrent Weekly Nedaplatin or Cisplatin With IMRT in NPC Patients
Brief Title: Weekly Cisplatin or Nedaplatin Concurrent With Intensity-modulated Radiation Therapy in Nasopharyngeal Carcinoma
Acronym: NPC-RCT-WCRT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: He Xia (Other)
Responsible Party: Sponsor-Investigator, He Xia, Jiangsu Cancer Hospital, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JiangsuCIH
Record Dates: First submitted 2014-11-19; First posted 2014-11-25 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — nedaplatin; Cisplatin

ARMS (4):
- Low dose cisplatin arm (Active Comparator): concurrent chemotherapy: cisplatin 20mg/m2,weekly,for 6 cycles during radiotherapy
  Interventions: Drug: Cisplatin
- High dose cisplatin arm (Active Comparator): concurrent chemotherapy: cisplatin 30mg/m2,weekly,for 6 cycles during radiotherapy
  Interventions: Drug: Cisplatin
- Low dose nedaplatin arm (Experimental): concurrent chemotherapy: nedaplatin 20mg/m2,weekly,for 6 cycles during radiotherapy
  Interventions: Drug: Nedaplatin
- High dose nedaplatin arm (Experimental): concurrent chemotherapy: nedaplatin 30mg/m2,weekly,for 6 cycles during radiotherapy
  Interventions: Drug: Nedaplatin

INTERVENTIONS:
Drug: Nedaplatin — Nedaplatin combine with IMRT
  Other Names: NDP
  Arms: High dose nedaplatin arm; Low dose nedaplatin arm
Drug: Cisplatin — Cisplatin combine with IMRT
  Other Names: PDD; DDP; CDDP
  Arms: High dose cisplatin arm; Low dose cisplatin arm

SUMMARY:
This is a randomized Phase III study to evaluate efficancy of weekly cisplatin or nedaplatin concurrent with Intensity-modulated radiation therapy in Nasopharyngeal Carcinoma (NPC).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed untreated NPC patients
* T1-2N1-3M0 or T3-4NxM0
* 18-70 years old
* with MRI examinations
* ECOG ≤ 2
* With written consent

Exclusion Criteria:

* With a second cancer
* Pregnancy
* With other severe diseases (blood,liver ,kidney or heart diseases)
* Could not be staged properly
* Without written consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2 years
Progress-free survival | 2 years

SECONDARY OUTCOMES:
Tumor response | radiotherapy in 2 week、4 week、7 week
Overall survival | 2 years